CLINICAL TRIAL: NCT06377865
Title: Thyroid Function , HbA1c in Relation to Ferritin Level in Adullt Patient e B Thalassemia
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Demiana Adel Aziz, resident, Assiut University
Other Study IDs: endocrine dis & B thalassemia
Record Dates: First submitted 2024-03-19; First posted 2024-04-22 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-03

CONDITIONS: B Thalassemia
MeSH Terms: conditions — beta-Thalassemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: Beta thalassemia ( major)
- 2: Beta thalassemia (intermediate)

SUMMARY:
to evaluate thyroid function ,HbA1C,&lipid profile in thalassemic patient to correlate thyroid function , Hba1c , lipid profile e ferritin level in thalassemic patient

DETAILED DESCRIPTION:
B-Thalassemia major (b-TM) is a hereditary ،anemia resulting from defects in the production of b-globin chains and is one of the most common genetic disorders worldwide.

The clinical classification of thalassemias is currently widely applied in clinical practice related to transfusion requirements Transfusion-dependent thalassemia (TDT) is defined as a condition where patients cannot produce adequate hemoglobin to survive without blood transfusion. Non-transfusion-dependent thalassemia (NTDT) is a descriptive term for patients who do not require regular lifelong transfusions. They may require intermittent or frequent transfusions in certain clinical situations.

Patients with β-thalassemia intermedia have symptoms in between carriers and those with β-thalassemia major.

Endocrine complications are the commonest among BTM patients and the attributing factor is iron deposition in endocrine organs due to frequent blood transfusions along with suboptimal iron chelation. Thus, keeping an iron level within the useful and safe range is critical since a low amount can cause anemia, while a high level can cause tissue damage Background pathophysiologic mechanism leading to DM in TM is unclear; some regard the iron induced pancreas cytotoxicity as the most significant contributor, a new hypothesis suggests the exhaustion of beta pancreatic cells subsequent to a chronic period of hyperinsulinemia .There are 5% of thalassemia patients develop clinical hypothyroidism that requires treatment, a bigger number of them develop subclinical compensated hypothyroidism with normal T3 and T4 levels but high TSH serum levels.

The TDT is also associated with altered lipid levels because of oxidative stress that can lead to early atherosclerosis, adding to the morbidity and even early mortality.

ELIGIBILITY:
Inclusion Criteria:

* patient aged18 and older
* both gender
* patient diagnosed B thalassemia major
* patient diagnosed B thalassemia intermediate

Exclusion Criteria:

* thalaasemia trait
* age less than 18
* type 1 D.M
* pt known thyroid &recive tttt

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patient aged18 and older ,both gender. patient diagnosed B thalassemia major &intermediate
Sampling Method: Non-Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Thyroid function ,Hba1c in relation to ferritin level in adult patients with beta thalassemia | 24 month
  HbA1c in thalassemia major versus intermediate

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa Haridy, Prof, Principal Investigator — Yes

REFERENCES:
- [Background] Inati A, Noureldine MA, Mansour A, Abbas HA. Endocrine and bone complications in beta-thalassemia intermedia: current understanding and treatment. Biomed Res Int. 2015;2015:813098. doi: 10.1155/2015/813098. Epub 2015 Mar 5. PMID 25834825
- [Background] Ray S, Saikia D, Vashisht Y, Sharma S, Meena RK, Kumar M. Dyslipidemia and atherogenic indexes in children with transfusion-dependent thalassemia. Hematol Transfus Cell Ther. 2024 Oct-Dec;46(4):345-351. doi: 10.1016/j.htct.2023.02.006. Epub 2023 Apr 22. PMID 37147168
- [Background] Chatterjee R, Bajoria R. New concept in natural history and management of diabetes mellitus in thalassemia major. Hemoglobin. 2009;33 Suppl 1:S127-30. doi: 10.3109/09553000903347880. PMID 20001615
- [Background] Mariotti S, Pigliaru F, Cocco MC, Spiga A, Vaquer S, Lai ME. beta-thalassemia and thyroid failure: is there a role for thyroid autoimmunity? Pediatr Endocrinol Rev. 2011 Mar;8 Suppl 2:307-9. PMID 21705983
- [Background] Fernandes JL. MRI for Iron Overload in Thalassemia. Hematol Oncol Clin North Am. 2018 Apr;32(2):277-295. doi: 10.1016/j.hoc.2017.11.012. PMID 29458732
- [Background] Vichinsky E. Non-transfusion-dependent thalassemia and thalassemia intermedia: epidemiology, complications, and management. Curr Med Res Opin. 2016;32(1):191-204. doi: 10.1185/03007995.2015.1110128. Epub 2015 Nov 25. PMID 26479125
- [Background] Kattamis A, Forni GL, Aydinok Y, Viprakasit V. Changing patterns in the epidemiology of beta-thalassemia. Eur J Haematol. 2020 Dec;105(6):692-703. doi: 10.1111/ejh.13512. Epub 2020 Sep 21. PMID 32886826
- [Background] Musallam KM, Cappellini MD, Viprakasit V, Kattamis A, Rivella S, Taher AT. Revisiting the non-transfusion-dependent (NTDT) vs. transfusion-dependent (TDT) thalassemia classification 10 years later. Am J Hematol. 2021 Feb 1;96(2):E54-E56. doi: 10.1002/ajh.26056. Epub 2020 Dec 9. No abstract available. PMID 33219703